CLINICAL TRIAL: NCT01068379
Title: Randomized Clinical Trial of Cryotherapy Versus Postoperative Laser Photocoagulation for Retinopexy in Scleral Buckle Surgery
Brief Title: Clinical Trial of Cryotherapy Versus Postoperative Laser Photocoagulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Rodrigo Pessoa Cavalcante Lira, Unicamp
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cryo laser
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: rhegmatogenous retinal detachment; cryopexy; photocoagulation
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryopexy (Experimental): the cryopexy was performed by placement of a normal spherical probe under the bucklings, around the break. The number of cryo applications was limited in number of 3. Freezing was stopped at the beginning of retinal whitening.
  Interventions: Procedure: criopexy
- laser photocoagulation 4 weeks after (Experimental): Laser-retinopexy was performed after proper positioning the patients; laser energy was delivered by depressing a foot pedal. Short burn duration (0.1 seconds) and low (300-miliWatts) power settings were used initially, and both the burn duration and power were gradually increased as determined by observation.
  Interventions: Procedure: laser

INTERVENTIONS:
Procedure: criopexy — he cryopexy was performed by placement of a normal spherical probe under the bucklings, around the break. The number of cryo applications was limited in number of 3. Freezing was stopped at the beginning of retinal whitening.
  Arms: Cryopexy
Procedure: laser — Laser-retinopexy was performed after proper positioning the patients; laser energy was delivered by depressing a foot pedal. Short burn duration (0.1 seconds) and low (300-miliWatts) power settings were used initially, and both the burn duration and power were gradually increased as determined by observation.
  Arms: laser photocoagulation 4 weeks after

SUMMARY:
The purpose of this randomized clinical trial was to compare reattachment rates among patients with rhegmatogenous retinal detachment who underwent scleral buckle surgery with retinopexy by cryotherapy versus postoperative (one month) laser photocoagulation.

DETAILED DESCRIPTION:
The purpose of this randomized clinical trial was to compare reattachment rates, visual acuity results and epiretinal membrane formation among patients with rhegmatogenous retinal detachment who underwent scleral buckle surgery with retinopexy by cryotherapy versus postoperative (one month) laser photocoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Primary rhegmatogenous retinal detachment with a single peripherical retinal break. All patients were phakic, under eighteen years old, with partial posterior vitreous detachment, visual loss or symptoms (floaters and photopsia) less than 30 days

Exclusion Criteria:

* No patient had a retinal break greater than 30 degrees, or retinal detachment larger than two quadrants, history of uveitis or infectious retinopathy, presence of Proliferative vitreoretinopathy (B or C), macular disease, glaucoma, hemoglobinopathy, diabetic retinopathy, and history of trauma or previous vitreoretinal surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was one week reattachment rate | 1 week

REFERENCES:
- [Derived] Lira RP, Takasaka I, Arieta CE, Nascimento MA, Caldato R, Panetta H. Cryotherapy vs laser photocoagulation in scleral buckle surgery: A randomized clinical trial. Arch Ophthalmol. 2010 Dec;128(12):1519-22. doi: 10.1001/archophthalmol.2010.271. PMID 21149772